CLINICAL TRIAL: NCT06882577
Title: Heart Evaluation of Acute Ischemic Stroke With Reperfusion Therapy
Acronym: HEART
Status: Recruiting | Type: Observational
Sponsor: Soochow University (Other)
Responsible Party: Principal Investigator, Jianqiang Ni, Clinical Professor, The First Affiliated Hospital of Soochow University
Other Study IDs: 2025PJ160
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; heart; Reperfusion Therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — anticoagulant peripheral blood, serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart Evaluation of Acute ischemic stroke with Reperfusion Therapy: Acute ischemic stroke within 24 h after onset of stroke-related symptoms.
  Interventions: Other: observational only- no intervention

INTERVENTIONS:
Other: observational only- no intervention — observational only- no intervention

SUMMARY:
Heart Evaluation of Acute ischemic stroke with Reperfusion Therapy (HEART) is a single-center observational registry evaluating the heart of patients hospitalized for acute ischemic stroke with reperfusion therapy.

This registry aims to establish quantified risk stratification and prognostic models, as well as suggest effective diagnostic and therapeutic strategies.

DETAILED DESCRIPTION:
There is growing evidence pointing to close interactions between acute ischemic stroke (AIS) and heart diseases. Heart diseases may lead to AIS (heart-to-brain interactions), with many cardiac conditions have been proposed as potential sources of cerebral embolism, and studies have also shown that AIS can induce cardiac injury (brain-to-heart interactions), namely Stroke-Heart Syndrome. In addition, due to the commonly shared risk factors, AIS patients had a significantly higher frequency of coexisting prior known or unknown coronary heart disease (brain-and-heart interactions). These heart problems not only add complexity to the etiological diagnosis but also account for a great proportionate mortality in AIS patients with reperfusion therapy, which is the most effective treatment method for AIS. The interconnected and coexisting properties of AIS and heart diseases requires a comprehensive scheme to evaluate, prevent, and treat patients.

Heart Evaluation of Acute ischemic stroke with Reperfusion Therapy (HEART) is a single-center observational registry evaluating the heart of patients hospitalized for acute ischemic stroke with reperfusion therapy.

This registry aims to establish quantified risk stratification and prognostic models, as well as suggest effective diagnostic and therapeutic strategies.

The clinical, laboratory and imaging information will be collected at the baseline. During an estimated 3-year follow-up, the diagnostic or monitoring procedures, treatment, functional status and new vascular events will be recorded by web-based patients' self-reports, investigators' regular telephone visits.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by patient
2. Age ≥ 18 years
3. Acute ischemic stroke (with matching brain lesion on MR imaging)
4. Enrolment within 24 h after onset of stroke-related symptoms.

Exclusion Criteria:

1. Pregnancy and / or breast-feeding.
2. Participation in an interventional study.
3. Patients refuse to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients within 24 h after onset of stroke-related symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Cardiovascular Events | 1 year
  cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina

SECONDARY OUTCOMES:
Rate of Major Adverse Cardiovascular Events | 90 days
  ardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina
Functional Outcome | 90 days
  Percentage of patients with modified Rankin Scale (mRS) scores (minimum 0 and maximum 5) 3 to 5, who are considered to be disabled.
Rate of Ischemic Stroke | 1 year
  fatal and nonfatal ischemic stroke.
Rate of Acute Coronary Syndrome | 1 year
  fatal and nonfatal myocardial infarction and unstable angina
Rate of Cardiovascular Mortality | 1 year
  any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death
Time to First Major Adverse Cardiovascular Event | 3 years
  from the date of enrollment until the date of first documented cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction or unstable angina, whichever comes first, assessed up to 3 years
Time to First Ischemic Stroke | 3 years
  from the date of enrollment until the date of first documented ischemic stroke, assessed up to 3 years
Rate of Major Adverse Cardiovascular Events | 3 years
  cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina
Rate of Ischemic Stroke | 3 years
  fatal and nonfatal ischemic stroke
Rate of Acute Coronary Syndrome | 3 years
  fatal and nonfatal myocardial infarction and unstable angina
Rate of Cardiovascular Mortality | 3 years
  any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided